CLINICAL TRIAL: NCT06176911
Title: A Multicenter, Open-label, Randomized, Controlled, Phase 2 Trial Comparing the Efficacy and Safety of Teriflunomide Plus Danazol in Patients With Steroid-resistant/Relapse ITP
Brief Title: The Combination of Teriflunomide and Danazol for Steroid-resistant/Relapse Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Luhe Hospital (Other); Chinese PLA General Hospital (Other); Navy General Hospital, Beijing (Other); Beijing Hospital (Other Government); Beijing Friendship Hospital (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); China-Japan Friendship Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-TFITP-01
Record Dates: First submitted 2023-12-06; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Immune Thrombocytopenia
Keywords: Teriflunomide; Danazol
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — teriflunomide; Danazol

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned at a 1:1 ratio to receive teriflunomide plus danazol or danazol. Each group requires 62 patients (considering a 10% drop-off).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teriflunomide plus danazol (Experimental): Oral teriflunomide was given at a starting dose of 7 mg once daily and danazol was given at a dose of 200mg twice daily for 24 weeks. Treatment was discontinued if very severe or life-threatening adverse events developed or at the patient's request.
  Interventions: Drug: Teriflunomide; Drug: Danazol
- Danazol (Active Comparator): Danazol was given at a dose of 200 mg twice a day for 24 weeks. Treatment was discontinued if very severe or life-threatening adverse events developed or at the patient's request.
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: Teriflunomide — Starting dose of 7 mg once daily. Dose adjustments are made throughout the study based on individual platelet counts.
  Other Names: AUBAGIO
  Arms: Teriflunomide plus danazol
Drug: Danazol — 200 mg twice daily.

SUMMARY:
To compare the efficacy and safety of teriflunomide plus danazol versus danazol in patients with steroid-resistant/relapse ITP

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, controlled trial of 124 adult patients with steroid-resistant/relapse ITP in China. Patients were randomized to receive either experimental teriflunomide plus danazol or active comparator danazol monotherapy. Treatment was discontinued if very severe or life-threatening adverse events developed or at the patient's request.

ELIGIBILITY:
Inclusion Criteria:

1. Primary immune thrombocytopenia (ITP) confirmed by excluding other supervened causes of thrombocytopenia;
2. Patients who did not achieve a sustained response to treatment with full-dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid tapering or after its discontinuation;
3. Patients with a platelet count <30,000/μL or a platelet count <50,000/μL with bleeding manifestations at the enrollment;
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Secondary immune thrombocytopenia (e.g. patients with HIV, HCV, Helicobacter pylori infection, or patients with confirmed autoimmune disease);
2. Active or a history of malignancy;
3. Pre-existing acute or chronic liver disease, or serum alanine aminotransferase (ALT) greater than two times the upper limit of normal (ULN);
4. Pregnancy or lactation;
5. Current or recent (< 4 weeks prior to screening) clinically serious viral, bacterial, fungal, or parasitic infection;
6. Active or chronic viral infection from hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV);
7. Have evidence of active tuberculosis (TB), or have previously had evidence of active TB and did not receive appropriate and documented treatment, or have had household contact with a person with active TB and did not receive appropriate and documented prophylaxis for TB;
8. Have experienced a clinically significant thrombotic event within 24 weeks of screening or are on anticoagulants and in the opinion of the investigator are not well controlled;
9. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Sustained response | From the start of study treatment (Day 1) to the end of week 24
  Platelet count over 30,000/μL and at least a 2-fold increase of the baseline count in the absence of bleeding and rescue therapy for at least four of the six visits between weeks 19 and 24.

SECONDARY OUTCOMES:
Overall response | From the start of study treatment (Day 1) to the end of week 24
  Complete response (CR) was defined as platelet count over 100,000/μL and absence of bleeding. Response (R) was defined as platelet count over 30,000/μL and at least a 2-fold increase of the baseline count and absence of bleeding.
Time to response | From the start of study treatment (Day 1) to the end of week 24
  The time from treatment initiation to achieve a CR or a R.
Duration of response | From the start of study treatment (Day 1) to the end of week 24
  The time from the achievement of a complete response or a partial response to the loss of response.
Initial response | From the start of study treatment (Day 1) up to week 4 of treatment
  The number of participants with achievement of CR or R at 4 weeks.
Bleeding events | From the start of study treatment (Day 1) to the end of week 24
  Clinically significant bleeding was assessed using the World Health Organization (WHO) bleeding scale.
Adverse events | From the start of study treatment (Day 1) to the end of week 24
  Adverse events (AEs) were reported and graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Health-related quality of life (HRQoL) | From the start of study treatment (Day 1) to the end of week 24
  ITP-PAQ was used to assess the Health-Related Quality of Life (HRQoL) before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University Institute of Hematology, Peking University People's Hospital
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China